CLINICAL TRIAL: NCT06725186
Title: Improving Emotion Dysregulation and Interpersonal Conflict Among Families of Adolescents With ADHD
Brief Title: Regulating Emotions Like An eXpert Among Adolescents With ADHD
Acronym: RELAX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-1281
Record Dates: First submitted 2024-12-05; First posted 2024-12-10 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2024-12

CONDITIONS: RELAX Telehealth Intervention; Psychoeducational Waitlist Control; EMI Smartphone App Pilot
Keywords: ADHD; telehealth; emotion regulation; family conflict; parenting
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Emotional Regulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RELAX Intervention (Experimental): group-based RELAX telehealth intervention
  Interventions: Behavioral: RELAX
- Psychoeducational Waitlist Control (Active Comparator): The psychoeducational component will consist of infographics regarding emotion regulation strategies and managing interpersonal conflict.
  Interventions: Behavioral: Psychoeducational Materials

INTERVENTIONS:
Behavioral: RELAX — The RELAX intervention is a social-emotional intervention consisting of 8 weekly, 1.5 hr sessions and a booster session 1 month and 6 months after the completion of RELAX. During the first 60 minutes of RELAX sessions, parents and adolescents meet separately; during the last 30 minutes combined parent-adolescent discussion and problem-solving activities take place. RELAX is structured such that parents learn emotion regulation/coping skills the week prior to them being taught to the adolescents. Group sessions will involve both didactics and discussion of topics including psychoeducation, basic cognitive/behavioral principles, emotional awareness, emotion regulation strategies, parent emotion socialization practices, coping skills, conflict management strategies, and communication skills.
  Arms: RELAX Intervention
Behavioral: Psychoeducational Materials — Infographics with information on emotion regulation development, emotion regulation strategies, and strategies for managing interpersonal conflict, including when different strategies are more or less effective will be provided to participants via email.
  Arms: Psychoeducational Waitlist Control

SUMMARY:
This study consists of a randomized controlled trial assessing the acceptability, feasibility, and efficacy of the RELAX (Regulating Emotions Like An eXpert) Intervention. Following randomization, 30 families will receive the RELAX intervention and 30 families will receive psychoeducational materials as part of a control condition. Additionally, 10 families from the RELAX condition will participate in a pilot study and focus groups to give feedback on developed smartphone apps to support skill use during and following completion of RELAX.

DETAILED DESCRIPTION:
This study seeks to quantify the efficacy of the telehealth RELAX intervention (n = 30) relative to a psychoeducational waitlist control (PWL; n = 30) through a RCT. The psychoeducational component will consist of infographics for parents and adolescents regarding ER strategies, parent emotion socialization, and managing interpersonal conflict. Participants will be 60 adolescents with ADHD in middle or high school (ages 11-16) who display moderate to severe emotion dysregulation as measured by the Difficulties in Emotion Regulation Scale, and a primary caregiver. Adolescents will have an estimated verbal IQ ≥ 80, as indicated by the Wechsler Intelligence Scale for Children, Fifth Edition Verbal Comprehension Index, with no evidence of severe developmental delay. All participants must be proficient in English. Adolescents may have comorbid conditions, so the sample will represent real-world adolescents with ADHD.

Ten families who complete the RELAX intervention will be asked to participate in the ecological momentary intervention (EMI) pilot study which will assess the developed EMI procedure's acceptability, appropriateness, and feasibility of using smartphone apps to practice the skills learned during RELAX both during the original 8 weekly sessions and throughout the 6 month follow-up period using Likert-ratings. Additionally, they will be asked if they are interested in accessing the mobile apps for a 4-week period to continue practicing the skills learned in RELAX and to provide more in-depth feedback on the app to the research team via a 1-hour focus group.

ELIGIBILITY:
Inclusion Criteria:

* child with ADHD in middle or high school at time of study entry
* child has an estimated verbal IQ >=80 based on the Wechsler Intelligence Scale for Children, Fifth Edition Verbal Comprehension Index
* child has no evidence of severe developmental delay either from genetic origins (e.g., Down Syndrome) or complications during pregnancy/birth (e.g., infection, micropremature)
* participating parent/legal guardian has custody/medical decision making of the child
* family uses English as one of their primary languages (i.e., able to participate in study visits and intervention conducted in English)

Exclusion Criteria:

* child not diagnosed with ADHD as confirmed by prior documented diagnosis and/or current comprehensive ADHD assessment as part of intake visit
* having a child outside of the eligible age range of 11-16 at time of study enrollment
* participating parent not having legal custody of the child
* having parents or children who are not fluent in English
* having a child with a severe developmental delay either from genetic origins (e.g., Down Syndrome) or complications from pregnancy/birth (e.g., infection, micro-premature)
* child has an IQ < 70.

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Difficulties in Emotion Regulation Scale - Short Form (DERS-SF) | From enrollment to the 6-month follow-up period.
  The DERS-SF will be used to assess emotion regulation problems (e.g., poor emotion awareness, poor emotion clarity, non-acceptance of emotions, poor access to emotion regulation strategies). The DERS will be completed at all timepoints by both parents and adolescents, with parents completing ratings for themselves and for their adolescents. The 18 DERS items are rated on a 5-point scale ranging from 1 - Almost Never (0-10%) to 5 - Almost Always (91-100%) and the total score represents a sum across items (with 3 items reversed score; range = 18-90) such that higher scores indicate greater dysregulation.
Cognitive Emotion Regulation Questionnaire (CERQ) | From enrollment to the 6-month follow-up period.
  The CERQ is a 36-item scale designed to evaluate cognitive aspects of emotion regulation or cognitive coping strategies (e.g., self-blame, rumination, putting into perspective, positive reappraisal, acceptance). Parents and adolescents are asked to rate what they generally think when they experience negative or unpleasant events on a 5-point Likert scale ranging from 1 (almost never) to 5 (almost always). Each subscale consists of 4 items. Of the 4 items included in a scale a sum score is made (simple straight count), which can range from 4 (never used) to 20 (often used cognitive coping strategy). Not more than 1 of the 4 items included in a scale may be 'missing'. In that case, the 'missing' score is replaced by the average of the three remaining scores. In this manner, even in the case of a missing value, a scale score ranging from 4 to 20 is obtained, with higher scores indicating more often using that particular cognitive coping strategy.
Observed Parent Emotion Socialization Strategies | From enrollment to the 6-month follow-up period.
  The Conflict Discussion Task will be coded for parent emotion socialization in response to adolescents' distress through seven possible reactions: emotion-focused (i.e., empathy and validation), problem-focused (i.e., targeting the stressor itself with questions and advice), minimizing (i.e., dismissing the affect as unimportant), punitive (i.e., blaming the adolescent for the affect); magnifying (i.e., intensifying adolescents' affect), autonomy-inhibiting (i.e., interfering with adolescents' independence in dealing with their affect), and facilitative engagement (i.e., general sensitivity and responsiveness to adolescents' attempts to discuss affect). Responses are coded on a scale representing an (1) absence, (2) minimal, (3) moderate, or (4) strong presence of the behavior reflected. These codes will be collapsed into supportive (emotion-focused, problem-focused, facilitative engagement) and non-supportive (minimizing, punitive, magnifying, autonomy-inhibiting) responses.
Conflict Behavior Questionnaire (CBQ) | From enrollment to the 6-month follow-up period.
  The CBQ consists of 20 true-false questions regarding how well parent and adolescents get along, get angry at each other, and behaviors that occur during arguments. The CBQ total score ranges from 0-20 with higher scores indicating more parent-adolescent conflict.
Coping with Children's Negative Emotions Scale (CCNES) - Adolescent Version - | From enrollment to the 6-month follow-up period.
  Parent and adolescent report on the CCNES Adolescent Version will be collected to assess changes in parent emotion socialization. The CCNES-Adolescent consists of 9 hypothetical situations, each with 6 possible responses for how parents would react rated on a 7-point Likert scale ranging from 1 - Very Unlikely to 7 - Very Likely. These 6 response types each become a subscale (distress, punitive, expressive encouragement, emotion-focused, problem-focused, and minimization), with each subscale score representing the mean rating across the 9 items. These 6 subscales can be further collapsed into supportive (expressive encouragement, emotion-focused, problem-focused) and non-supportive (distress, punitive, minimization) responses, with higher scores indicating a greater likelihood a parent will use that particular response type.

SECONDARY OUTCOMES:
Center for Epidemiological Studies Depression Scale for Children (CES-DC) | From enrollment to the 6-month follow-up period.
  Adolescent self-report of their depression symptoms will be collected using the CES-DC. The CES-DC consists of 20 items assessing depression symptoms rated on a 4-point scale (0 = Not At All, 4 = A Lot). The CES-DC total score represents the sum across the 20 items, with possible scores ranging from 0 to 60. Higher CES-DC scores indicate increasing levels of depression.
Screen for Child Anxiety Related Emotional Disorders (SCARED) | From enrollment to the 6-month follow-up period.
  Adolescent self-report on the SCARED will be used to measure adolescent anxiety symptoms. The SCARED consists of 41 items rated on a 3-point scale (0 = Not True or Hardly Ever True, 2 = Very True or Often True). The SCARED measures overall anxiety symptoms, Panic Disorder, Generalized Anxiety Disorder, Separation Anxiety, Social Anxiety, and School Avoidance. Higher scores on each subscale represent more anxiety symptoms. The overall anxiety total score will be used in the current study; scores can range from 0-82, with higher scores indicating more anxiety symptoms and a total score of ≥ 25 indicating the possible presence of an Anxiety Disorder.
Proactive and Reactive Aggression Measure (PRAM) | From enrollment to the 6-month follow-up period.
  The PRAM will be used to measure adolescent self-reported proactive and reactive aggression. The PRAM consists of 6 items that differentiate between reactive aggression (3 items; e.g., "When I have been teased or threatened I get angry easily and strike back") and proactive aggression (3 items; e.g., "I threaten or bully others in order to get my way."). Items are anchored on a 5-point scale (1 = never, 5 = almost always). The two subscales range from 3 - 15 points; the total aggression score ranges from 6 - 30 points, with higher scores indicating the presence of more aggression in the adolescent.
Self-Injurious Thoughts and Behaviors | From enrollment to the 6-month follow-up period.
  Adolescent report on a questionnaire developed from the Self-Injurious Thoughts and Behaviors Interview will be used to assess suicide ideation, plans, gestures, and attempts, and non-suicidal self-injury. First, adolescents are asked if they have ever had thoughts of killing themselves. If they answer yes, they are asked how old they were the first time they had thoughts of killing themself, how often (# of weeks in last year) they have had such thoughts, and the last time they had thoughts of killing themself. Next, they are asked if they ever wish they were dead followed by if they ever made a plan to kill themself; if they respond yes to either or both, the same 3 follow-up questions are asked for each. Then they are asked if they have ever attempted suicide. If they answer yes, they are asked how old they were at the first attempt, how many attempts they have had, the last attempt, and the method used for the attempts. Finally, injury resulting from attempts or NSSI is assessed.
Vanderbilt ADHD Rating Scale (VARS) | From enrollment to the 6-month follow-up period.
  The VARS will be used to assess parent report of ADHD, ODD, and CD symptoms, and social and academic impairment. The VARS consists of 40 symptom items (18 ADHD, 8 ODD, 14 CD) rated on a 4-point scale ranging from 0 - Never to 3 - Very Often. Any item endorsed as happening Often or Very Often is counted as a clinical symptom for that disorder, with the symptom count for each disorder being used and higher values indicating more symptom severity. Finally, 8 impairment items are asked on which the parents rate how much various areas (School Performance; Relationships with Parents, Siblings, Peers; Participation in Organized Activities) problems for the child on a 5-point scale ranging from 1 - Excellent Performance to 5 - Problematic. A total impairment score can be calculated by summing the 8 items (range = 8 - 40), with higher scores indicating more impairment in each domain.
Homework Performance Questionnaire (HPQ) | From enrollment to the 6-month follow-up period.
  Academic performance will be measured using parent report on the HPQ. The HPQ items are on a 7-point Likert scale ranging from 0 (Never/Rarely, 0-10% of the time) to 6 (Almost Always/Always, 91% to 100% of the time). Percentages indicate how often a behavior occurs, with items worded in the positive such that 91-100% means the adolescent does that behavior consistently well. Thus, higher scores indicate less impairment.
Depression Anxiety Stress Scales - 21 item (DASS-21) | From enrollment to the 6-month follow-up period.
  The DASS-21 will be used to assess parents' report of their own depression, anxiety, and stress symptoms, given evidence that parent depression and stress is related to child emotional and behavioral outcomes and ratings of child behavior. The 21 items are rated on a 4-point scale ranging from 0 - Did not apply to me at all to 3 - Applied to me very much, or most of the time, indicating how often over the past week they have experienced the various symptoms. Each subscale (depression, anxiety, stress) consists of 7 items (range = 0 - 21), with the DASS-21 total score ranging from 0 - 63, with higher scores indicating more severe internalizing symptoms (scores of 28+ are considered extremely severe on this measure).
Alabama Parenting Questionnaire - Short Form (APQ-9) | From enrollment to the 6-month follow-up period.
  The APQ-9 will be used to assess changes in parent and adolescent report on global parenting behaviors. Each of the 9 items are rated on a 5-point scale ranging from Never (1) to Always (5). The scores for each of the three subscales are added together to create three subscale scores: Positive parenting (Items 1, 6 and 7), Inconsistent discipline (Items 2, 4, and 9), and Poor supervision (items 3, 5, 8), which values ranging from 3 - 15 for each subscale and higher values indicating a greater likelihood that these parenting behaviors typically occur in their home.

CONTACTS AND LOCATIONS:
Overall Officials: Rosanna Breaux, PhD, Principal Investigator — Virginia Polytechnic Institute and State University
Locations (1):
- Child Study Center, Blacksburg, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Breaux, R., Shroff, D. M., Cash, A. R., Swanson, C. S., Carlton, C., Bertollo, J. R., & Dahiya, A. V. (2023). Telehealth delivery of the RELAX intervention for families of adolescents diagnosed with ADHD: Preliminary treatment outcomes and evidence of acceptability and feasibility. Evidence-Based Practice in Child & Adolescent Mental Health, 8, 24-38. doi: 10.1080/23794925.2021.1970053
- See also: CALMER Lab Website Description of the RELAX Intervention — https://www.calmerlab.com/the-relax-intervention